CLINICAL TRIAL: NCT01958710
Title: Outcome After Surgical Treatment or Bronchial Embolisation in Aspergilloma of the Lung: a Single Center Experience.
Brief Title: Outcome After Treatment of Pulmonary Aspergilloma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, Datamanager Thoracic Surgery, University Hospital, Gasthuisberg
Other Study IDs: ASPERLEU
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Fungal Diseases
Keywords: Catheterization, Bronchial; Pneumonectomy; Lobectomy; Thoracoplasty
MeSH Terms: conditions — Lung Diseases, Fungal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Embolisation: (preoperative) embolisation of the bronchial circulation
- Surgery: Any surgically treated patient with a functional lung resection (at least wedge resection)

SUMMARY:
Retrospective analysis of surgery and/or bronchial embolisation for pulmonary aspergilloma.

DETAILED DESCRIPTION:
A retrospective chart analysis, based on the search results from a thoracic surgery database and an interventional radiology database. Outcome analysis of all surgically treated patients for a confirmed invasive aspergilloma. Comparisson with (preoperative) embolisation of the bronchial circulation.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven Aspergilloma of the lung

Exclusion Criteria:

* Treatment limited to the use of systemic antifungal agents

Ages: 1 Year to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the database with following interventions will be screened for invasive aspergilloma in the final resection specimen:
  Aspergilloma Fungal disease Lung bleeding Destroyed lung Empyema of the lung
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
survival after treatment | 10 years
  estimated 10 yaer survival after treatment for pulmonary aspergilloma

SECONDARY OUTCOMES:
post treatment survival | 90 days
  survival status at 90 days after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Decaluwé, MD, Principal Investigator — UZ Leuven - dept. Thoracic Surgery; Laurence Bertrand, MSc, Principal Investigator — Katholic University Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium